CLINICAL TRIAL: NCT07173881
Title: Effect of Consumption of a Dairy Product Designed for Pregnant and Lactating Women on the Composition of Human Milk. A Quasi-experimental Study in a Vulnerable Population
Brief Title: Effect of a Dairy Product for Pregnant and Lactating Women on the Composition of Human Milk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Desarrollo e Investigaciones Pediátricas Prof. Dr. Fernando E. Viteri (Other)
Collaborators: Hospital Interzonal de Agudos General San Martín (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UCTH 2025
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy
Keywords: human milk; vulnerable population; pregnancy; nutritional supplements; esencial fatty acids; micronutrients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Super 1.000 Mamá (Experimental): Pregnant women who will consume a fortified powdered dairy product formulated and designed specifically for this population during pregnancy and the first month postpartum.
  Interventions: Dietary Supplement: Fortified powder milk
- Sham Comparator: No milk consumption (No Intervention): Breastfeeding women who have not consumed SMM until the first month postpartum

INTERVENTIONS:
Dietary Supplement: Fortified powder milk — Super 1.000 Mamá It's made up of milk with added vegetable oils, fish oil, carbohydrates from corn, prebiotic fiber (inulin), vitamins, and minerals, with specifically defined proportions. It has medium energy content, is balanced in protein, fats, and carbohydrates, and provides a significant content of both polyunsaturated fatty acids, such as omega-6, and omega-3, and the added docosahexaenoic acid, as recommended by international organizations. The reconstituted 200 ml serving delivers between 20 and 40% of the Daily Reference Intake in critical nutrients for this particular group of people, which include minerals such as calcium, iron, zinc, iodine, and vitamins such as A, D, C, B12 and folic acid. The rest of the vitamins, and minerals are also at the same level, allowing those who consume it to incorporate a large amount of nutrients regularly. Addvance SA, an SME dairy company from the Province of Santa Fe, will carry out the production of this milk.
  Arms: Experimental: Super 1.000 Mamá

SUMMARY:
Vulnerable populations, who have deficient diets, may produce human milk (HML) that is not adequate in all nutrients, and this will have consequences on the growth and development of the child. In 2021, at IDIP, a specific milk product for pregnant and lactating women, Super Mil Mamá ( SMM, whole milk powder fortified with multiple vitamins, minerals, and DHA ) was designed and developed as part of a key strategy to incorporate into public policies for the first 1000 days of life. However, the potential benefits of this product have not yet been evaluated at the population level. The main objective is to evaluate the effect of the consumption of a milk product (SMM) designed for pregnant women on maternal nutritional status and the composition of human milk at one month postpartum.

Specific objectives include:

To compare the concentrations of DHA, Vitamins A, E, and D, Iron, Iodine, Zinc, and Calcium in human milk at one month postpartum of mothers who consumed SSM or not.

To compare the concentrations of DHA, Vitamins A, E, D and Zinc in blood and the nutritional status of maternal iron between mothers who consumed SSM and those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Intervention group: Pregnant women over 18 years of age who undergo prenatal care during gestational weeks (GW) 28 ± 1 at the Maternal Nutrition Clinic of the H.I.G.A. "San Martín" in La Plata, and who regularly consume milk, will be included.
* Control group: Women over 18 years of age who attend their child's first checkup before the first month of life at the Maternal Clinic of the IDIP Health Observatory, and who exclusively breastfeed their children, will be included.

Exclusion Criteria:

* Women who have had multiple pregnancies and/or women with malabsorption diseases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Breast milk DHA concentration | Time Frame: breast milk DHA concentration will be assessed at one month postpartum.
  Description: concentration of DHA in breast milk expressed as a percentage of DHA with respect to the total fatty acids contained in the analyzed sample
Mother Zinc concentration | Mother Zinc concentration will be assessed at one month postpartum
  Zinc concentration in mother serum expressed in mg/dl
mother Vit E concentration | Mother's serum α-tocopherol concentration will be assessed at one month postpartum
  α-tocopherol concentration in mother serum expressed in μmol/L
Mother Vit A concentration | Mother's Vit A concentration will be assessed at one month postpartum
  Retinol concentration in mother serum expressed in μmol/L
Mother red blood cell DHA concentration | Mother's serum DHA concentration will be assessed at one month postpartum
  Concentration of DHA in mother's red blood cell expressed as a percentage of DHA with respect to the total fatty acids contained in the analyzed sample
Mother hemoglobin concentration | Mother's hemoglobin concentration will be assessed one month postpartum
  hemoglobin concentration in mother serum expressed in g/dL
Breast milk Vitamin A concentration | Breast milk Vitamin A concentration will be assessed at one month postpartum
  Retinol concentration in breast milk expressed in μmol/L and μg/g fat contained in the analyzed sample
Breast milk Vitamin E concentration | Breast milk Vitamin E concentration will be assessed at one month postpartum
  α-tocopherol concentration in breast milk expressed in μmol/L and μg/g fat contained in the analyzed sample
Breast milk Vitamin D concentration | Breast milk Vitamin D concentration will be assessed at one month postpartum
  25-hidroxi vitamin D concentration in breast milk expressed in ng/ml
Breast milk Zinc concentration | Breast milk Zinc concentration will be assessed at one month postpartum
  Zinc concentration in breast milk expressed in mg/dl
Breast milk Calcium concentration | Breast milk Calcium concentration will be assessed at one month postpartum
  Calcium concentration in breast milk expressed in mg/dl
Breast milk Iron concentration | Breast milk Iron concentration will be assessed at one month postpartum
  Iron concentration in breast milk expressed in mg/dl
Breast milk Iodine concentration | Breast milk Iodine concentration will be assessed at one month postpartum
  Iodine concentration in breast milk expressed in mg/dl
Mother serum ferritin concentration | Mother's serum ferritin concentration will be assessed at one month postpartum
  ferritin concentration in mother serum expressed in ng/ml
mother Vit D concentration | mother Vit D concentration will be assessed at one month postpartum
  25-hidroxi vitamin D concentration in mother serum expressed in ng/ml

CONTACTS AND LOCATIONS:
Locations (2):
- Argentina (2):
  - Hospital Interzonal de Agudos General San Martín, La Plata, Buenos Aires
  - Instituto de Desarrollo e Investigaciones Pediátricas (IDIP) - HIAEP Sor María Ludovica, La Plata, Buenos Aires